CLINICAL TRIAL: NCT01582477
Title: Evaluation of the Safety and Efficacy of EXPAREL When Administered by Infiltration Into the Transversus Abdominis Plane (TAP) for Prolonged Postsurgical Analgesia in Subjects Undergoing Robot-assisted Laparoscopic Prostatectomy
Brief Title: TAP-patients With Robotic Assisted Lap Prostatectomy
Acronym: TAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA402S23B701
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Postsurgical Pain; Analgesia; Prostatectomy
Keywords: TAP, robot-assisted prostatectomy
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EXPAREL 20 mL (undiluted) (Experimental): 20 mL (266 mg) undiluted EXPAREL with 133 mg infiltrated on each the right and left side of the abdomen.
  Interventions: Drug: EXPAREL 20 mL
- EXPAREL 40 mL (diluted) (Active Comparator): 20 mL (266 mg) EXPAREL diluted with an equal volume of preservative-free 0.9% normal saline to a total of 40 mL and infiltrated equally to the right and left side of the abdomen.
  Interventions: Drug: EXPAREL 40 mL

INTERVENTIONS:
Drug: EXPAREL 20 mL — EXPAREL 266 mg (undiluted)
  Other Names: bupivacaine liposome injectable suspension
  Arms: EXPAREL 20 mL (undiluted)
Drug: EXPAREL 40 mL — EXPAREL 266 mg diluted with preservative-free 0.9% normal saline to 40 mL.
  Other Names: bupivacaine liposome injectable suspension
  Arms: EXPAREL 40 mL (diluted)

SUMMARY:
The purpose of the study is to assess the safety and efficacy of EXPAREL when administered via infiltration into the transversus abdominis plane (TAP) to prolonged postsurgical analgesia in men undergoing robot-assisted laparoscopic prostatectomy.

DETAILED DESCRIPTION:
Assess the safety and efficacy of EXPAREL when administered via infiltration into the transversus abdominis plane (TAP) to provide prolonged postsurgical analgesia in men undergoing robot-assisted laparoscopic prostatectomy. The primary endpoint is the duration of abdominal analgesia from the infiltration into the TAP as measured by the time to the subject's first postsurgical opioid administration.

ELIGIBILITY:
Inclusion Criteria:

* male subjects, aged 18-75.
* American Society of Anesthesiology (ASA) physical status 1-3.
* Undergoing robot-assisted laparoscopic prostatectomy performed by a single surgeon (Ingolf Tuerk, MD).
* Subjects must be physically and mentally able to participate in the study and complete all study assessments.
* Subjects must be able to give fully informed consent to participate in this study after demonstrating a good understanding of the risks and benefits of the TAP infiltration.

Exclusion Criteria:

* Demonstrated hypersensitivity or idiosyncratic reactions to amide-type local anesthetics.
* Inability to tolerate oxycodone with acetaminophen (e.g. Percocet).
* Any subject whose anatomy or surgical procedure in the opinion of the Investigator might preclude the potential successful performance of a TAP.
* Any subject who in the opinion of the Investigator might be harmed or be a poor candidate for participation in the study.
* Subjects who have received any investigational drug within 30 days prior to study drug administration or planned administration of another investigational product or procedure during their participation in this study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sternlicht, MD, Principal Investigator — Steward St. Elizabeth's
Locations (1):
- Steward St. Elizabeth's, Brighton, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- EXPAREL 20 mL: Group receiving EXPAREL 20 mL
- EXPAREL 40 mL: Group receiving EXPAREL 40 mL
Period: Overall Study
Arm/Group | EXPAREL 20 mL | EXPAREL 40 mL
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EXPAREL 20 mL | EXPAREL 40 mL | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 9 | 15
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (7.24) | 61.7 (7.01) | 61.2 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: The Duration of Abdominal Analgesia From Infiltration Into the TAP
Time Frame: First postsurgical administration of an opioid
Population: Per protocol
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | EXPAREL 20 mL | EXPAREL 40 mL
Number analyzed (Participants) | 12 | 12
hours | 0.39 [0.27 to 0.60] | 0.44 [0.40 to 0.58]

2. Secondary Outcome: Subject Reported Postsurgical Pain
Description: 11-point numeric rating scale (NRS) (0-10, where 0=no pain, 10=worst possible pain)
Time Frame: 1, 2, 6, 12, 24, 48, 72, 96 hours and 10 days after TAP
Population: Number analyzed in one or more rows differs from overall number analyzed in the instances that participant did not complete the assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXPAREL 20 mL | EXPAREL 40 mL
Number analyzed (Participants) | 12 | 12
units on a scale
  1 hour after TAP | 4.4 (2.57) | 5.3 (2.35)
  2 hours after TAP | 3.1 (1.5) | 3.9 (2.15)
  6 hours after TAP: number analyzed (Participants) | 11 | 11
  6 hours after TAP | 2.4 (1.57) | 3.0 (2.10)
  12 hours after TAP: number analyzed (Participants) | 10 | 11
  12 hours after TAP | 2.5 (2.12) | 2.2 (1.60)
  24 hours after TAP | 1.8 (1.75) | 2.5 (1.68)
  48 hours after TAP | 2.0 (1.54) | 2.5 (2.61)
  72 hours after TAP | 1.8 (1.64) | 1.9 (1.83)
  96 hours after TAP | 1.1 (1.08) | 1.7 (2.06)
  Day 10 after TAP: number analyzed (Participants) | 10 | 11
  Day 10 after TAP | 0.00 (0.00) | 1.0 (1.55)

3. Secondary Outcome: Physician/Healthcare Professional Assessed Postsurgical Pain
Description: 11-point NRS (0-10, 0=no pain, 10=worst possible pain)
Time Frame: 1, 2, 6, 12, 24 hours after TAP
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXPAREL 20 mL | EXPAREL 40 mL
Number analyzed (Participants) | 12 | 12
units on a scale
  1 hour after TAP | 4.2 (2.33) | 5.3 (2.35)
  2 hours after TAP | 2.9 (1.56) | 3.9 (2.15)
  6 hours after TAP: number analyzed (Participants) | 11 | 11
  6 hours after TAP | 2.4 (1.57) | 3.0 (2.10)
  12 hours after TAP: number analyzed (Participants) | 10 | 11
  12 hours after TAP | 2.6 (2.07) | 2.2 (1.33)
  24 hours after TAP | 1.8 (1.75) | 2.5 (1.68)

4. Secondary Outcome: Total Postsurgical Oxycodone/Acetaminophen Consumption From Hospital Discharge Through Hour 96.
Description: Number of pills
Time Frame: 48, 72, 96 hours
Measure: Mean (Standard Deviation); unit: Number of tablets
Arm/Group | EXPAREL 20 mL | EXPAREL 40 mL
Number analyzed (Participants) | 12 | 12
Number of tablets
  48 hours | 1.9 (2.11) | 2.2 (2.12)
  72 hours | 2.8 (3.21) | 3.4 (3.75)
  96 hours | 3.7 (4.25) | 4.8 (5.33)

5. Secondary Outcome: Incidence of Prespecified Opioid-related Adverse Events
Description: Number of subjects
Time Frame: Until hospital discharge order was written, anticipated at 24 hours.
Measure: Number; unit: Number of subjects
Arm/Group | EXPAREL 20 mL | EXPAREL 40 mL
Number analyzed (Participants) | 12 | 12
Number of subjects | 0 | 0

6. Secondary Outcome: Overall Rating of Subject Satisfaction With Postsurgical Pain Control
Description: Mean of subject satisfaction offered on a 5-point Likert scale (1 = extremely dissatisfied, 2 = dissatisfied, 3 = neither satisfied nor dissatisfied, 4 = satisfied, 5 = extremely satisfied)
Time Frame: 24 hours, 72 hours, and day 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | EXPAREL 20 mL | EXPAREL 40 mL
Number analyzed (Participants) | 12 | 12
Participants
  24 hours- satisfied | 4 | 5
  24 hours- extremely satisfied | 8 | 7
  72 hours - satisfied: number analyzed (Participants) | 11 | 11
  72 hours - satisfied | 4 | 4
  72 hours - extremely satisfied: number analyzed (Participants) | 11 | 11
  72 hours - extremely satisfied | 7 | 7
  Day 10 - satisfied: number analyzed (Participants) | 11 | 11
  Day 10 - satisfied | 3 | 4
  Day 10- extremely satisfied: number analyzed (Participants) | 11 | 11
  Day 10- extremely satisfied | 8 | 7

ADVERSE EVENTS:
Arm/Group | EXPAREL 20 mL | EXPAREL 40 mL
Serious Adverse Events (participants affected / at risk) | 3/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXPAREL 20 mL (N=12) | EXPAREL 40 mL (N=12)
Post-procedural Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXPAREL 20 mL (N=12) | EXPAREL 40 mL (N=12)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No